CLINICAL TRIAL: NCT04029337
Title: An Early Feasibility Study of the HighLife 28mm Trans-Septal Transcatheter Mitral Valve Replacement System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HighLife SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-2019-01
Record Dates: First submitted 2019-07-20; First posted 2019-07-23 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Transcatheter Mitral Valve Replacement (Experimental): HighLife TMVR System is a novel and innovative approach developed as an alternative treatment for severe MR when medical treatment is maximal and surgical interventions not possible or at high risk. The HighLife TMVR system is composed of a Transcatheter Mitral Valve (TMV), a sub-annular implant (SAI), and their delivery systems and loading tools.
  Interventions: Device: Transcatheter Mitral Valve Replacement

INTERVENTIONS:
Device: Transcatheter Mitral Valve Replacement — Minimally invasive transcatheter mitral valve implantation using the HighLife™ TMVR system

SUMMARY:
Study to evaluate the feasibility, safety and performance of the HighLife trans-septal Transcatheter Mitral Valve in patients with moderate-severe and severe mitral regurgitation who are at high risk for surgical treatment.

DETAILED DESCRIPTION:
Protocol Title:

An Early Feasibility Study of the HighLife 28mm Transcatheter Trans-Septal Mitral Valve Replacement System

Protocol # HL-2019-01, ver. 5.0

Phase: United States Early Feasibility Study

Investigational Devices:

The HighLife 28mm Trans-Septal Mitral Valve and its delivery systems. These devices compose the HighLife Trans-septal Mitral Valve Replacement (TSMVR) System.

* Size 28 mm TMV (CLARITY valve)
* Size 28 mm TMV-L (CLARITY large annulus valve/ LAV)

Intended Use: The HighLife TSMVR system is intended for the trans-septal access percutaneous mitral valve replacement in patients suffering from symptomatic moderate-severe or severe mitral regurgitation (MR) due to primary (degenerative) or secondary (functional) abnormality of the mitral valve.

Device Description:

The HighLife TSMVR system is composed of a Trans-Septal (Mitral Valve (TSMV), a sub-annular implant (SAI), and their delivery systems and accessories. The TMV is a 28 mm mitral bioprosthesis made of a self-expanding Nitinol frame covered with polyester graft and supporting bovine pericardium leaflets. The bioprosthesis is used in conjunction with the Sub-Annular Implant (SAI), comprising a ring (made of polycarbonate urethane (PCU), nitinol, gold markers and polyester (Dacron) to be placed around the mitral valve apparatus to stabilize the position of the mitral valve implant.

Design: A single arm, prospective, multicenter, non-randomized and open-labelled study.

Purpose: The purpose of the study is to evaluate the feasibility, safety and performance of the HighLife 28mm Trans-septal Mitral Valve Replacement (TSMVR) system in NYHA Class ≥ II-IV patients with moderate-severe or severe mitral regurgitation who are at high risk for surgical treatment or deemed more appropriate to receive transcatheter mitral valve replacement than to receive conventional mitral valve surgery according to the local multidisciplinary Heart Team.

Objectives: Primary objectives are to evaluate the feasibility, safety and performance of the HighLife 28mm TSMVR system at 30 days. Secondary objectives are to evaluate long term safety and performance of the HighLife TSMVR system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe mitral regurgitation
* New York Heart Association (NYHA) Functional Class II, III or ambulatory IV.
* Patient is under maximally tolerated GDMT (incl. CRT) for at least 3 months
* Multidisciplinary Heart Team consensus that the patient is inoperable or at high-risk for surgical repair/replacement due to significant co-morbid conditions
* Multidisciplinary Heart Team consensus that the patient is not a suitable candidate for other approved percutaneous repair therapy due to anatomical or medical conditions
* Patient meets the anatomical criteria for HighLife valve sizing as determined by CT and TEE

Main Exclusion Criteria:

* Mitral stenosis
* Rheumatic valve disease
* Severe calcifications of the mitral annulus and/or mitral leaflets
* Prior surgical or interventional treatment of the mitral valve
* Unsuitable anatomy for the transapical access
* Unsuitable anatomy of the aorta and ilio-femoral vessels for the transfemoral access
* Untreated clinically significant coronary artery disease requiring revascularization
* LVEF < 30%
* LVEDD > 70mm
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Hypertrophic Obstructive Cardiomyopathy (HOCM)
* Any surgical or interventional procedure (including PCI) done in the past 30 days prior to procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Freedom of major adverse events | at 30 days post procedure
  including:
  * All-cause mortality
  * Myocardial infarction or coronary ischemia requiring PCI or CABG
  * Major stroke
  * Life-threatening bleeding (MVARC scale)
  * Major access and vascular complications
  * Stage 2 or 3 acute kidney injury (includes dialysis)
  * Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention
  * Severe hypotension, heart failure or respiratory failure requiring intravenous pressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for ≥ 48H
Continued intended performance of the HighLife™ bioprosthesis | at 30 days post procedure
  defined as the reduction of mitral regurgitation (MR) to either optimal (0+ to trace) or acceptable (reduced by at least 1 grade from baseline with no more than 2+ MR) without significant mitral stenosis (post-procedure EOA ≥ 1.5 cm2 with a transmitral gradient < 5mmHg) and with no greater than mild (1+) paravalvular MR (and without associated hemolysis)

SECONDARY OUTCOMES:
Technical success | immediately after procedure
  defined as alive patient at exit from procedure room, with all of the following:
  * Successful access, delivery and retrieval of the HighLife delivery systems
  * Deployment and correct positioning of the HighLife bioprosthesis
  * Freedom of additional emergency surgery or re-intervention related to the device or access procedure

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Tucson Medical Center, Tucson, Arizona
  - Los Robles Regional Medical Center, Los Angeles, California
  - Piedmont Heart, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minneapolis Heart, Minneapolis, Minnesota
  - Montefiore Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Hospital, Houston, Texas
  - Chippenham Hospital Richmond, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No